CLINICAL TRIAL: NCT03724006
Title: Impact Assessment of a Psychoeducational Intervention in Quality of Life of Parents With Children With Congenital Heart Defects
Brief Title: Impact of Psychoeducation in Quality of Life of Parents With Children With Congenital Heart Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Unidade Autónoma de Gestão da Mulher e Criança do Centro Hospitalar Universitário de São João (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PPeCHD; SFRH/BD/123908/2016 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-07

CONDITIONS: Congenital Heart Defects
Keywords: Congenital Heart Defects; Diagnosis; Parents; Quality of Life; Education
MeSH Terms: conditions — Heart Defects, Congenital; Disease

STUDY DESIGN:
Intervention Model Description: Parents will be divided in 2 study groups: INTERVENTION group (I) and CONTROL group (C).
  Group I will receive a psychoeducational intervention in addition to the usual routines of the Service. Group C will receive the usual routines of the Service. The intervention will be performed as soon as possible after inclusion in the study.
  Participants will be evaluated in 3 moments: M1 beginning of the study; M2 4 weeks after the intervention (I) or after enrollment (C) and M3 16 weeks after intervention/enrollment. The primary outcome will be parental QoL, which will be evaluated through the WHOQOL-Bref. The family impact and the perception of positive contributions will be secondary outcomes. These outcome variables will be assessed by the Impact on Family Scale and the Positive Contributions Scale - Kansas Inventory of Parental Perceptions, respectively. A semi-structured interview will be performed after all quantitative data have been collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION group (I) (Experimental): Group I will be composed by parents of children with the diagnosis of CHD who will receive a psychoeducational intervention plus usual routines of the Service.
  Interventions: Behavioral: Psychoeducational intervention
- CONTROL group (C) (No Intervention): Group C will be composed by parents of children with the diagnosis of CHD who will receive the usual routines of the Service. After completing the data collection, the possibility of receiving the psychoeducational intervention under study will be offered to this group.

INTERVENTIONS:
Behavioral: Psychoeducational intervention — The intervention, prepared by a multidisciplinary team, will consist of two 90 minutes collective sessions (max. 8 families). Sessions will consist of lectures, group discussion and relaxation. The program includes content on the effects of a diagnosis of a congenital anomaly on a child in the parents and in the family, stages of mourning, adaptation process, coping strategies, legislative framework and social protection. This is a non-specific intervention for CHD, where the main focus is the diagnosis of a congenital anomaly.
  In second session, written support material will be distributed. Participants will be asked to practice relaxation in the next 4 weeks.
  Arms: INTERVENTION group (I)

SUMMARY:
Congenital heart defects (CHD) are the most common congenital malformations. Despite the progress made in the last decades in diagnosis and treatment, CHD continues to be associated with significant morbidity and mortality. Several studies have shown a reduction in the quality of life (QoL) of parents of children with CHD, which may affect children too. The main research aim is to assess and to understand the impact of a psychoeducational intervention in QoL of parents with newborns with CHD.

We are including parents of inpatient newborns in Neonatal Intensive Care Unit (NICU) of UAG da Mulher e Criança - Centro Hospitalar Universitário de São João (CHUSJ) with the diagnosis of non-syndromic CHD, between March 2019 and February 2020. We also included parents of newborns born at CHUSJ with the diagnosis of non-syndromic CHD, not admited in NICU, between September 2019 and February 2020. The inclusion criteria are: I) parents of newborns (up to 28 days) with the diagnosis of non- syndromic CHD; II) newborns hospitalized in CHUSJ; III) parents aged ≥ 18 years. Parents of newborns with other important co-morbidities associated with CHD and those who do not have good understanding and expression in Portuguese will be excluded.

Parents will be divided in 2 study groups: INTERVENTION group (I) and CONTROL group (C). Group I will receive a psychoeducational intervention in addition to the usual routines of the Service. Group C will receive the usual routines of the Service. The psychoeducational intervention, which consists of 2 sessions lasting 90 minutes each one, will be performed as soon as possible after inclusion in the study. Participants will be evaluated in three moments: M1 beginning of the study; M2 4 weeks after the intervention (I) or after enrollment (C) and M3 16 weeks after intervention/enrollment. The primary outcome will be parental QoL, which will be evaluated through the World Health Organization Quality of Life-Bref (WHOQOL-Bref). The family impact and the perception of positive contributions will be secondary outcomes. These outcome variables will be assessed by the Impact on Family Scale and the Positive Contributions Scale - Kansas Inventory of Parental Perceptions, respectively. A semi-structured interview will be performed after all quantitative data have been collected.

The authors expect to find an increase of QoL and positive contributions and a decrease of family impact in the intervention group comparatively to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Parents of newborns (up to 28 days) with the diagnosis of non-syndromic CHD;
* Newborns hospitalized in CHUSJ;
* Parents aged ≥ 18 years.

Exclusion Criteria:

* Parents of newborns with other important comorbidities associated with CHD;
* Parents who do not have good understanding and expression in Portuguese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Changes on parental QoL | INTERVENTION group - M1: baseline (beginning of the study); M2: 4 weeks after the intervention and M3: 16 weeks after intervention. CONTROL group - M1: baseline; M2: 4 weeks after enrollment and M3: 16 weeks after enrollment.
  Changes on parental quality of life assessed through World Health Organization Quality of Life-Bref (WHOQOL-Bref). The WHOQOL-Bref instrument is composed by 26 items, which are organized in 4 specific domains: Physical (7 items), Psychological (6 items), Social Relationships (3 items), Environment (8 items) and a general QoL facet (2 items). All items are quoted from 1 to 5. Three items, related to questions posed negatively (Q3, Q4 and Q26), must be reversed (the calculation implies the subtraction of their value to six units). The results are transformed on a scale of 0 to 100. Each domain score is computed through the formula: [(sum of all items - number of items) / (4x number of items)] x 100. Higher scores correspond to better quality of life.

SECONDARY OUTCOMES:
Changes on family impact | INTERVENTION group - M1: baseline (beginning of the study); M2: 4 weeks after the intervention and M3: 16 weeks after intervention. CONTROL group - M1: baseline; M2 4 weeks after enrollment and M3 16 weeks after enrollment.
  Changes on family impact assessed through Revised Impact on Family Scale. Impact on Family Scale evaluates the parents' perception of the impact of the child's chronic health condition in family life. Revised Impact on Family Scale contains 15 items. It is a unidimensional scale that scores overall family impact. This score results from sum of all item responses. The result ranges from 15 to 60. Higher scores are indicative of perceived higher family impact associated with child's health condition.
Changes on perception positive contributions | INTERVENTION group - M1: baseline ( beginning of the study); M2: 4 weeks after the intervention and M3: 16 weeks after intervention. CONTROL group - M1: baseline; M2: 4 weeks after enrollment and M3: 16 weeks after enrollment.
  Changes on perception positive contributions assessed through Positive Contributions Scale - Kansas Inventory of Parental Perceptions. The Portuguese version of the Positive Contributions Scale - Kansas Inventory of Parental Perceptions is composed by 43 items that assessed 6 dimensions/subscales: 1) Source of Personal Growth and Future Consciousness; 2) Source of Learning Out of Experience; 3) Source of Acceptance and Family Cohesion; 4) Source of Happiness and Affection; 5) Source of Spirituality and 6) Source of Social Network Expansion. The scores of the subscales are computed by the average of the items that composes them. Higher scores indicate a perception of greater positive contributions in the different dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Rodrigues, MD, Principal Investigator — Centro de Investigação em Tecnologias e Serviços de Saúde; Faculdade de Medicina da Universidade do Porto; Centro Hospitalar Universitário de São João; Maria Emília Areias, PhD, Study Chair — Instituto Universitário de Ciências da Saúde da Cooperativa do Ensino Superior, Politécnico e Universitário; Unidade de Investigação e Desenvolvimento Cardiovascular do Porto; José Carlos Areias, PhD, Study Chair — Faculdade de Medicina da Universidade do Porto; Unidade de Investigação e Desenvolvimento Cardiovascular do Porto; Pedro Pereira Rodrigues, PhD, Study Chair — Centro de Investigação em Tecnologias e Serviços de Saúde; Departamento de Medicina da Comunidade Informação e Decisão em Saúde; Faculdade de Medicina da Universidade do Porto; Luís Filipe Azevedo, PhD, Study Chair — Centro de Investigação em Tecnologias e Serviços de Saúde; Departamento de Medicina da Comunidade Informação e Decisão em Saúde; Faculdade de Medicina da Universidade do Porto
Locations (1):
- Centro Hospitalar Universitário de São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigues MG, Rodrigues JD, Moreira JA, Clemente F, Dias CC, Azevedo LF, Rodrigues PP, Areias JC, Areias ME. A randomized controlled trial to assess the impact of psychoeducation on the quality of life of parents with children with congenital heart defects-Quantitative component. Child Care Health Dev. 2024 Jan;50(1):e13199. doi: 10.1111/cch.13199. Epub 2023 Nov 15. PMID 37967565
- See also: Assessment methods and levels of quality of life of parents with children with congenital abnormalities - systematic review and meta-analysis. — https://www.crd.york.ac.uk/prospero/display_record.php?RecordID=62271
- See also: Psycho-educational interventions effectiveness to improve the quality of life of parents of children with congenital abnormalities - systematic review and meta-analysis - systematic review and meta-analysis. — https://www.crd.york.ac.uk/prospero/display_record.php?RecordID=79534
- See also: Impact of psycho-educational interventions in quality of life of parents of children with chronic diseases - systematic review and meta-analysis. — https://www.crd.york.ac.uk/prospero/display_record.php?RecordID=92135